CLINICAL TRIAL: NCT00902187
Title: An Open-Label, Randomized, Single-Dose, Two-Way Crossover Bioequivalence Study Of 4 Mg Fesoterodine Extended-Release Tablets (Toviaz™), Manufactured At Zwickau Versus Vega Baja, In Healthy Subjects.
Brief Title: A Bioequivalence Study Of 4 Mg Fesoterodine Extended-Release Tablets (Toviaz™) In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0221081
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Treatment of Overactive Bladder
Keywords: Bioequivalence
MeSH Terms: interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference (Other): fesoterodine (Toviaz™ 4 mg) tablet manufactured at Zwickau (Reference)
  Interventions: Drug: Fesoterodine
- Test (Other): fesoterodine (Toviaz™ 4 mg) tablet manufactured at Vega Baja (Test)
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Fesoterodine — A fesoterodine extended-release tablet (ER) formulation once daily administration of 4 mg
  Other Names: Toviaz 4 mg
  Arms: Reference
Drug: Fesoterodine — A fesoterodine extended-release tablet (ER) formulation once daily administration of 4 mg
  Other Names: Toviaz 4 mg
  Arms: Test

SUMMARY:
To demonstrate bioequivalence of fesoterodine 4 mg tablets manufactured at Vega Baja, versus Zwickau.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Subjects with evidence or history of clinically significant urologic diseases
* A positive urine drug screen
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
AUCinf, AUClast, and Cmax of 5-HMT | 6 weeks

SECONDARY OUTCOMES:
Tmax and half-life of 5-HMT as data permit | 6 weeks
Safety laboratory tests and adverse events | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221081